CLINICAL TRIAL: NCT04228835
Title: Does ICG Fluorescence Cholangiography Identify Critical View of Safety Earlier in Laparoscopic Cholecystectomy: Results From a Randomized Controlled Study in University Malaya Medical Centre
Brief Title: Does ICG Fluorescence Cholangiography Identify Critical View of Safety Earlier in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Ummi Surgical Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Dr Koong Jun Kit, Senior Lecturer and Consultant Surgeon, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1001
Record Dates: First submitted 2019-11-27; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Cholelithiasis
Keywords: Symptomatic and Complicated Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Intervention Model Description: Patients are divided into two arms: ICG enhanced fluorescence cholangiography assisted laparoscopic cholecystectomy (ICGFC- LC) and conventional laparoscopic cholecystectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICGFC-LC (Experimental): ICG fluorescence cholangiography assisted laparoscopic cholecystectomy (ICGFC-LC) arm patients received intravenous bolus of 2.5mg of ICG before the induction of anaesthesia. Near infrared laparoscopic light camera was utilized intermittently during dissection of Calot's triangle until critical view of safety was achieved.
  Interventions: Diagnostic Test: Fluorescence Cholangiography
- Conventional LC (No Intervention): Conventional laparoscopic cholecystectomy (LC) arm patients underwent standard white light laparoscopic cholecystectomy without fluorescence cholangiography.

INTERVENTIONS:
Diagnostic Test: Fluorescence Cholangiography — Administration of ICG for fluorescence cholangiography
  Arms: ICGFC-LC

SUMMARY:
Achievement of critical view of safety (CVS) is recommended to reduce risk of hilar injury in laparoscopic cholecystectomy. Indocyanine green (ICG) fluorescence cholangiography, a novel technique of real time biliary visualization, is postulated to assist dissection during laparoscopic cholecystectomy (LC). However, its use in providing a faster and safer LC has yet to be established. The main objective of this study is to evaluate whether the use of ICG enhanced fluorescence cholangiography will help in earlier identification critical view of safety during LC.

DETAILED DESCRIPTION:
Indocyanine green (ICG) is excreted exclusively in the biliary system and emits fluorescence light when viewed using near infrared imaging. This enables extrahepatic biliary tree anatomy to be delineated during laparoscopic cholecystectomy.

Indocyanine green fluorescence cholangiography also enables earlier detection of cystic duct and common bile duct during laparoscopic cholecystectomy. This is reported in two studies which showed that cystic duct can be identified 11 minutes and 8.6 minutes earlier and common bile duct 10 and 11 minutes earlier than white light imaging.

To date, there is no data published on the use of fluorescent cholangiography in reducing operative time of identification of critical view of safety during laparoscopic cholecystectomy, which is an integral part of the surgery. Theoretically achievement of critical view of safety maybe facilitated by fluorescent cholangiography as this technique facilitates identification of biliary structures.

The primary objective of this study is to evaluate whether an earlier identification of CVS can be obtained by using ICG fluorescence cholangiography as an adjunct to conventional laparoscopic cholecystectomy versus conventional laparoscopic cholecystectomy. Secondary outcomes assessed are the presence of minor or major complications between this two groups.

Patients are randomly assigned into two arms; ICG fluorescence cholangiography assisted laparoscopic cholecystectomy (ICGFC- LC) and conventional laparoscopic cholecystectomy (LC), using a computer-generated block randomization. Patients in the ICGFC- LC group received intravenous bolus of 2.5mg of ICG before the induction of anaesthesia. All the surgeries are performed using standard four ports technique. Near infrared light camera by Karl Storz Endoscopy is used intermittently during dissection for the ICGFC-LC group.

Time to identification of CVS is defined by time of gallbladder retraction to time of establishment of critical view of safety. Critical view of safety is achieved when all the three criteria set by Strasberg is met. Mean time to identification of CVS in the two groups of patients were then compared. All patients are followed up for one month to identify any post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cholelithiasis for elective cholecystectomy
* American Society of Anaesthesiologist (ASA) classification of physical status I or II
* Normal kidney function
* Normal liver function

Exclusion Criteria:

* Liver cirrhosis
* Hepatits B or C
* Allergies to iodine or seafood

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Time to identification of critical view of safety | Time of surgery
  Compare time to identification of critical view of safety during laparoscopic cholecystectomy which is defined as time of gallbladder retraction until establishment of critical view of safety.

SECONDARY OUTCOMES:
Complications | up to 30 days post operative
  Compare rate of complications of laparoscopic cholecystectomy such as bile duct injury, major haemorrhage, intraabdominal collections and surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Jun Kit Koong, MS, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schols RM, Bouvy ND, van Dam RM, Masclee AA, Dejong CH, Stassen LP. Combined vascular and biliary fluorescence imaging in laparoscopic cholecystectomy. Surg Endosc. 2013 Dec;27(12):4511-7. doi: 10.1007/s00464-013-3100-7. Epub 2013 Jul 23. PMID 23877766
- [Background] van Dam DA, Ankersmit M, van de Ven P, van Rijswijk AS, Tuynman JB, Meijerink WJ. Comparing Near-Infrared Imaging with Indocyanine Green to Conventional Imaging During Laparoscopic Cholecystectomy: A Prospective Crossover Study. J Laparoendosc Adv Surg Tech A. 2015 Jun;25(6):486-92. doi: 10.1089/lap.2014.0248. Epub 2015 May 14. PMID 25974072
- [Derived] Koong JK, Ng GH, Ramayah K, Koh PS, Yoong BK. Early identification of the critical view of safety in laparoscopic cholecystectomy using indocyanine green fluorescence cholangiography: A randomised controlled study. Asian J Surg. 2021 Mar;44(3):537-543. doi: 10.1016/j.asjsur.2020.11.002. Epub 2020 Nov 19. PMID 33223453